CLINICAL TRIAL: NCT06518161
Title: Développement d'un Atlas Des Interactions hôte-microbiome Respiratoire Chez Des Volontaires Sains
Brief Title: Development of an Atlas of Respiratory Host-microbiome Interactions in Healthy Volunteers
Acronym: HEALTHY LUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC24_0007
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Healthy Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voluntary (Other): Subjects undergoing scheduled surgery in the operating room at Nantes University Hospital, requiring general anesthesia with placement of an endotracheal intubation tube for invasive mechanical ventilation.
  Interventions: Other: Voluntary

INTERVENTIONS:
Other: Voluntary — Subjects undergoing scheduled surgery in the operating room at Nantes University Hospital, requiring general anesthesia with placement of an endotracheal intubation tube for invasive mechanical ventilation.

SUMMARY:
The role of the pulmonary microbiome in the pathophysiology of lung disease is becoming increasingly well understood. Studies on murine models have highlighted the immunomodulatory and antibacterial activity of certain commensal bacteria, such as S. mitis, and have led to an understanding of their potential therapeutic impact. The investigators will therefore couple their analyses of the respiratory microbiome with an in-depth analysis of mucosal immunity. In particular, they will characterize immune cell types and frequencies using high-dimensional (spectral) flow cytometry and single cell RNA-sequencing. Finally, they will study the mediators exchanged between the microbiome and the host using proteomic and metabolomic analyses of respiratory fluids.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age from 18 to 70.
* Indication for scheduled general anesthesia with orotracheal intubation for non-thoracic, non-carcinological, non-septic surgical procedures such as prosthesis (knee or hip), spinal surgery, digestive hernia surgery, gall bladder surgery, maxillofacial surgery (non-exhaustive list).
* Membership of a social security scheme or beneficiary of such a scheme.
* Written informed consent.

Exclusion Criteria:

* Persons under guardianship or trusteeship.
* Pregnant or breast-feeding woman.
* Antibiotic treatment received within 28 days prior to surgery, regardless of the site of infection.
* Acute respiratory pathology within the last 28 days (pneumothorax, bronchitis or pneumonia including Covid).
* History of chronic respiratory disease (asthma, chronic obstructive pulmonary disease, emphysema, lung cancer, cystic fibrosis, etc.).
* Immunosuppression (cancer active or within the last 5 years, HIV, radio-chemotherapy within the last year, organ transplant).
* Chronic inflammatory disease (digestive, osteoarticular, neurological or cutaneous) requiring or having required specific treatment in the last 12 months.
* Type I or II diabetes.
* Steroid treatment within the last 30 days (regardless of dose or duration).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Atlas of host-microbiome interactions | 1 day
  Healthy respiratory metacluster

SECONDARY OUTCOMES:
Correlations between bacterial species | Day 1
  To define the link between the patient and the bacterial transcriptional activities
Correlations between bacterial species | Day 1
  To define the link between the patient and the bacterial composition
Correlations between cell populations | Day 1
  To define the link between the patient and the transcriptional clusters of cell populations
Correlations between metabolite concentrations | Day 1
  To define the link between the patient and the metabolite concentrations
Correlations between protein concentrations | Day 1
  To define the link between the patient and the protein concentrations
Correlations between host-microbiome interactions and quality of life scales | Day 1
  To define the link between the patient and different scales (MOCA, EPICES, modified MRC, NYHA, EQ5D-5L, SWLS, SF-36, HADS and BPI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided